CLINICAL TRIAL: NCT06223958
Title: A Phase 3, Multicenter, Double-Masked, Randomized, Parallel-Group Study to Evaluate the Efficacy and Safety of Intravitreal OTX-TKI (Axitinib Implant) in Subjects With Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: Study to Evaluate the Efficacy and Safety of Intravitreal OTX-TKI (Ocular Therapeutix) (Axitinib Implant) in Subjects With Neovascular Age-Related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Collaborators: Fortrea (Industry); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTX-TKI-2023-AMD-301; SOL-1 (Other: Ocular Therapeutix)
Record Dates: First submitted 2024-01-12; First posted 2024-01-25 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration; Tyrosine Kinase Inhibitor; OTX-TKI
MeSH Terms: interventions — Axitinib; aflibercept

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTX-TKI (axitinib implant) (Experimental)
  Interventions: Drug: OTX-TKI (axitinib implant)
- Control (Other)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: OTX-TKI (axitinib implant) — Intravitreal Injection of OTX-TKI (axitinib implant)
  Arms: OTX-TKI (axitinib implant)
Drug: Aflibercept — Injection of 2mg (0.05mL) of aflibercept
  Arms: Control

SUMMARY:
Study to Evaluate the Efficacy and Safety of Intravitreal OTX-TKI (axitinib implant) in Subjects with Neovascular Age-Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve for Neovascular Age-Related Macular Degeneration (nAMD) in either eye at screening.
* Are at least older than 50 years of age at Day 1.
* Have Best Corrected Visual Acuity (BCVA) of at least 84 Early Treatment Diabetic Retinopathy Study (ETDRS) letter score (approximate 20/20 Snellen equivalent) at Day 1; OR have an increase of at least 10 ETDRS letters of Best Corrected Visual Acuity (BCVA) from Screening (Visit 1) BCVA

Exclusion Criteria:

* Monocular subjects or a Best Corrected Visual Acuity (BCVA) score of 20/200 in fellow eye at screening.
* Have evidence of a scar, fibrosis, or atrophy of > 50% of the total lesion in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | Up to 36 Weeks
  Maintenance of visual acuity, defined as < 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters Best corrected visual acuity (BCVA) loss

OTHER OUTCOMES:
Incidence and severity of treatment emergent adverse events (AEs) | Up to 104 Weeks
  Changes Safety Outcomes from Baseline

CONTACTS AND LOCATIONS:
Locations (108):
- United States (97):
  - Associated Retina Consultants - Gilbert, Gilbert, Arizona
  - Associated Retina Consultants - Phoenix, Phoenix, Arizona
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - CA CRC California Retina Consultants, Bakersfield, California
  - The Retina Partners - Encino, Encino, California
  - Retina Consultants of Orange County - Fullerton, Fullerton, California
  - Atlantis Eyecare, Huntington Beach, California
  - Lakeside Vision Center - Irvine, Irvine, California
  - Retina-Vitreous Associates Medical Group - Los Angeles, Los Angeles, California
  - CA RCMG Retinal Consultants Medical Group, Inc., Modesto, California
  - Retina Sacramento MSO, LLC, Modesto, California
  - Kaiser Permanente Division of Research, Oakland, California
  - CA CRC California Retina Consultants, Oxnard, California
  - Stanford University School of Medicine, Byers Eye Institute, Palo Alto, California
  - Doheny Eye Center, Pasadena, California
  - AzulVision, Pasadena, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants (CRC) - Santa Barbara, Santa Barbara, California
  - Macula Retina Vitreous Center, Torrance, California
  - Bay Area Retina Associates, A Medical Group, Walnut Creek, California
  - Retina Consultants of Southern Colorado - Colorado Springs, Colorado Springs, Colorado
  - RSC Research, PLLC, Denver, Colorado
  - Colorado Retina Associates (CRA) - Lakewood, Lakewood, Colorado
  - Retina Group of New England, PC, Waterford, Connecticut
  - The Macula Center - Clearwater Office (Suncoast Retina Consultants, LLC), Clearwater, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - Speciality Retina Center, Deerfield Beach, Florida
  - Retina Group of Florida - Fort Lauderdale, Fort Lauderdale, Florida
  - Florida Retina Institute - Lake Mary, Lake Mary, Florida
  - Florida Retina Consultants - Lakeland, Lakeland, Florida
  - South Florida Retina Institute, Miami, Florida
  - Retina Specialty Institute - Pensacola, Pensacola, Florida
  - MedEye Associates - Miami, South Miami, Florida
  - Retina Vitreous Associates of Florida (RVA) - Saint Petersburg, St. Petersburg, Florida
  - Retina Vitreous Associates of Florida - Tampa, Tampa, Florida
  - Retina Associates of Florida LLC Tampa MacDill, Tampa, Florida
  - Southeast Retina Center, P.C. - Augusta, Augusta, Georgia
  - Illinois Eye and Ear Infirmary at UI Health UIC, Chicago, Illinois
  - Illinois Retina Associates, S.C. - Lincoln Park, Chicago, Illinois
  - University Retina and Macula Associates, P.C., Oak Forest, Illinois
  - Springfield Clinic, Springfield, Illinois
  - IN AVRUC Associated Vitreoretinal and Uveitis Consultants, Carmel, Indiana
  - Retina Partners Midwest, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Maine Eye Center - Marginal Way Campus, Portland, Maine
  - The Wilmer Eye Institute, Baltimore, Maryland
  - Mid Atlantic Retina Specialists - Hagerstown, Hagerstown, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Associated Retinal Consultants P.C. (ARC) - Royal Oak, Royal Oak, Michigan
  - Retina Consultants of Minnesota, Edina, Minnesota
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - Pepose Vision Institute, Chesterfield, Missouri
  - Retina Research Institute, LLC, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - The Retina Center Of New Jersey, LLC - Bloomfield, Bloomfield, New Jersey
  - Long Island Vitreoretinal Consultants (VRC) - Hauppauge, Hauppauge, New York
  - Retina-Vitreous Surgeons of Central New York, Liverpool, New York
  - NY LIVRC Long Island Vitreoretinal Consultants, Shirley, New York
  - Asheville Eye Associates (AEA) - Retinal Office, Asheville, North Carolina
  - Duke University Health System - Duke Eye Center Of North Durham, Durham, North Carolina
  - Retina Associates of Cleveland, Inc. - Beachwood, Beachwood, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Retina Associates of Cleveland, Inc. - Youngstown, Youngstown, Ohio
  - Erie Retina Research, Erie, Pennsylvania
  - Palmetto Retina Center, Aiken, South Carolina
  - Charleston Neuroscience Institute LLC - Beaufort, Beaufort, South Carolina
  - SC CNI Retina Consultants of Charleston, Beaufort, South Carolina
  - Charleston Neuroscience Institute LLC - Charleston, Charleston, South Carolina
  - Palmetto Retina Center, Florence, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Retina Consultants of Charleston - Mount Pleasant, Mt. Pleasant, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute (BHREI), Rapid City, South Dakota
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Charles Retina Institute PC, Germantown, Tennessee
  - Tennessee Retina, PC - Nashville - Centennial Professional Plaza Location, Nashville, Tennessee
  - West Texas Retina Consultants (WTRC) - Abilene (Ophthalmology Specialists of Texas, PA), Abilene, Texas
  - Texas Retina Associates (TRA) - Arlington, Arlington, Texas
  - Retina Consultants of Austin PA (RCA) - Central Austin, Austin, Texas
  - Austin Retina Associates, PLLC, Austin, Texas
  - Keystone Research, Austin, Texas
  - Retina Research Center (RRC), Austin, Texas
  - Retina Consultants of Texas Beaumont, Beaumont, Texas
  - Retina Group, Inc. d/b/a Retina Consultants of America (Retina Consultants of Texas), Bellaire, Texas
  - Star Vision Consultants, Burleson, Texas
  - Texas Retina Center, Houston, Texas
  - Retina Consultants of Texas - Katy, Katy, Texas
  - Medical Center Ophthalmology Associates (MCOA) - Northwest Clinic Location, San Antonio, Texas
  - Retinal Consultants of Texas - San Antonio Medical Center, San Antonio, Texas
  - TX RCTX Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Retina Associates of Utah, P.C - Intermountain Medical Center Location, Salt Lake City, Utah
  - Wagner Macula & Retina Center - Norfolk, VA Office, Norfolk, Virginia
  - Vistar Eye Center Vision and Surgery Specialists, Roanoke, Virginia
  - Eye Clinic of Wisconsin, Wausau, Wisconsin
- Argentina (10):
  - Buenos Aires Macula, Pilar, Buenos Aires
  - Centro Oftalmologico Dr. Charles S.A, Buenos Aires, Buenos Aires F.D.
  - Organizacion Medica de Investigacion OMI, Buenos Aires, Buenos Aires F.D.
  - Fundacion Zambrano - Cirugia Ocular, Buenos Aires, Buenos Aires F.D.
  - Instituto Oftalmologico de Alta Complejidad, Buenos Aires, Buenos Aires F.D.
  - Oftalmologia Global, Rosario, Santa Fe Province
  - Centro Privado de Ojos Romagosa SA, Córdoba
  - Oftar Mendoza Srl Centro Privado de Oftalmologia, Mendoza
  - Centrovision, Mendoza
  - Laser Vision Group, Santa Fe
- Emanuelli research and development, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided